CLINICAL TRIAL: NCT02291055
Title: Phase 1-2 Study of ADXS11-001 or MEDI4736 Alone or Combination In Previously Treated Locally Advanced or Metastatic Cervical or HPV+ Head & Neck Cancer
Brief Title: A Study of ADXS11-001 or MEDI4736 Alone or Combination In Cervical or Human Papillomavirus (HPV)+ Head & Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advaxis, Inc. (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADXS001-04
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Cervical Cancer; Cancer; Head and Neck Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms; Head and Neck Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 (Experimental): Participants with cervical cancer received MEDI4736 3 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 2 weeks (Q2W) at an infusion rate of approximately 60 minutes followed by ADXS11-001 1×10^9 CFU IV infusion every 4 weeks (Q4W) at an infusion rate of approximately 60 minutes. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
  Interventions: Drug: ADXS11-001; Drug: MEDI4736
- Part A Escalation (Cervical and Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (Experimental): Participants with cervical cancer and SCCHN received MEDI4736 10 mg/kg IV infusion Q2W at an infusion rate of approximately 60 minutes followed by ADXS11-001 1×10^9 CFU IV infusion Q4W at an infusion rate of approximately 60 minutes. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
  Interventions: Drug: ADXS11-001; Drug: MEDI4736
- Part A Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (Experimental): Participants with SCCHN received MEDI4736 10 mg/kg IV infusion Q2W at an infusion rate of approximately 60 minutes followed by ADXS11-001 1×10^9 CFU IV infusion Q4W at an infusion rate of approximately 60 minutes. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
  Interventions: Drug: ADXS11-001; Drug: MEDI4736
- Part B Expansion (Cervical): 10 mg/kg MEDI4736 (Experimental): Participants with cervical cancer received MEDI4736 10 mg/kg IV infusion Q2W at an infusion rate of approximately 60 minutes. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
  Interventions: Drug: MEDI4736
- Part B Expansion (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (Experimental): Participants with cervical cancer received MEDI4736 10 mg/kg IV infusion Q2W at an infusion rate of approximately 60 minutes followed by ADXS11-001 1×10^9 CFU IV infusion Q4W at an infusion rate of approximately 60 minutes. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
  Interventions: Drug: ADXS11-001; Drug: MEDI4736

INTERVENTIONS:
Drug: ADXS11-001
  Arms: Part A Escalation (Cervical and Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736; Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736; Part A Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736; Part B Expansion (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Drug: MEDI4736

SUMMARY:
This was a multicenter, open-label, 2-part randomized study of MEDI4736 administered as monotherapy or in combination with ADXS11-001 to participants with recurrent/persistent or metastatic squamous or non-squamous carcinoma of the cervix or metastatic human papillomaviruses (HPV)+ squamous cell carcinoma of the head and neck (SCCHN).

DETAILED DESCRIPTION:
The study was conducted in 2 parts Part A (dose-escalation and expansion) and Part B (expansion).

Part A:

Part A of the study was a Phase 1 dose escalation evaluation of the combination treatment of ADXS11-001 at a fixed dose of 1×10^9 colony-forming units (CFU) administered intravenously (IV) every 4 weeks (Q4W) and escalating doses of MEDI4736 (3 mg/kg and 10 mg/kg) administered IV every 2 weeks (Q2W) to determine the safety and tolerability of the combination and to identify a recommended Phase 2 dose (RP2D). Part A also included an expansion cohort of participants with metastatic SCCHN only. Once the RP2D was identified, the expansion cohort of Part A of the study were to commence.

Part B:

Part B of the study was a Phase 2 design in which participants who had failed at least 1 prior systemic treatment for their recurrent, persistent or metastatic cervical cancer were enrolled and randomized 1:1 to receive either MEDI4736 10 mg/kg alone or MEDI4736 10 mg/kg in combination with ADXS11-001 1×10^9 CFU.

ELIGIBILITY:
Inclusion Criteria:

1. Have histological diagnosis of SCCHN with confirmation of HPV positivity or squamous, non-squamous, adenosquamous, carcinoma or adenocarcinoma of the cervix which HPV positivity is not required
2. Have measurable and/or evaluable disease by response evaluation criteria in solid tumors (RECIST) 1.1
3. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Have adequate organ function defined by the protocol.

Exclusion Criteria:

1. Has any prior Grade ≥3 immune-related adverse event (irAE) while receiving immunotherapy, including anti-CTLA-4 treatment, or any unresolved irAE >Grade 1.
2. Has a diagnosis of immunodeficiency or is receiving any systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Day 1 of trial treatment.
3. Has any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for invasive malignancy within 2 years. Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
4. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
5. Has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screw(s), metal plate(s), bone graft(s), or other exogenous implant(s)). NOTE: More common devices and prosthetics which include arterial and venous stents, dental and breast implants, and venous access devices (e.g., Port-a-Cath or Mediport) are permitted. Sponsor must be contacted prior to consenting any subject who has any other device and/or implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Site, Los Angeles, California
  - Site, New Haven, Connecticut
  - Site, Jacksonville, Florida
  - Site, Miami, Florida
  - Site, Tampa, Florida
  - Site, Urbana, Illinois
  - Site, Lexington, Kentucky
  - Site, Baltimore, Maryland
  - Site, Detroit, Michigan
  - Site, Omaha, Nebraska
  - Site, Brooklyn, New York
  - Site, New York, New York
  - Site, Canton, Ohio
  - Site, Hilliard, Ohio
  - Site, Oklahoma City, Oklahoma
  - Site, Chattanooga, Tennessee
  - Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Slomovitz BM, Moore K, Vangala S, Parsi M, Sheerie S, John Heyburn J ,Posner M. Phase II study of durvalumab alone or in combination with ADXS11-001 (AXAL) in recurrent/persistent or metastatic cervical cancer. Annual Meeting on Women's Cancer. March 28-31, 2020. Toronto Canada.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in the United States.
Pre-assignment Details: Participants with a diagnosis of cervical cancer and human papillomavirus (HPV) positive squamous cell carcinoma of head and neck (SCCHN) were enrolled in the study.
Period: Overall Study
Arm/Group | Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A Escalation (Cervical and Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part A Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Started | 5 | 5 | 11 | 27 | 27
Completed | 0 | 0 | 3 | 0 | 0
Not Completed | 5 | 5 | 8 | 27 | 27
Not completed — Death | 2 | 2 | 5 | 8 | 12
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 5 | 10
Not completed — Progressive Disease | 0 | 0 | 1 | 4 | 2
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 5 | 1
Not completed — Other | 0 | 2 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Population included participants who received at least 1 dose of study drug.
Groups:
- Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736: Participants with cervical cancer received MEDI4736 3 mg/kg IV infusion Q2W at an infusion rate of approximately 60 minutes followed by ADXS11-001 1×10^9 CFU IV infusion Q4W at an infusion rate of approximately 60 minutes. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A Escalation (Cervical and Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part A Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Total
Number analyzed (Participants) | 5 | 5 | 11 | 27 | 27 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9 | 23 | 27 | 68
  >=65 years | 0 | 1 | 2 | 4 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 0 | 27 | 27 | 63
  Male | 0 | 1 | 11 | 0 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3 | 6 | 12
  Not Hispanic or Latino | 5 | 4 | 9 | 24 | 21 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 0 | 0 | 1 | 2
  Race: Black or African American | 1 | 0 | 1 | 5 | 3 | 10
  Race: White | 3 | 4 | 10 | 19 | 21 | 57
  Race: Other | 0 | 1 | 0 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) in Part A and Part B
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. Any worsening (ie, any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that was temporally associated with the use of the Sponsor's product, was also considered an AE. A serious adverse event (SAE) was any AE that: results in death; life threatening; resulted in or prolonged an existing inpatient hospitalization, persistent or significant disability/incapacity; congenital anomaly; a new cancer; associated with an overdose; another important medical event. Treatment emergent was defined as events with onset dates on or after the first dose of study medication and within 30 days following the last dose of study medication.
Time Frame: From first dose until 30 days after last dose (maximum duration: 98 weeks)
Population: All Treated Population.
Measure: Number; unit: participants
Arm/Group | Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A Escalation (Cervical and Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part A Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Number analyzed (Participants) | 5 | 5 | 11 | 27 | 27
participants
  TEAEs | 5 | 5 | 11 | 25 | 27
  TESAEs | 2 | 3 | 4 | 13 | 15

2. Primary Outcome: Progression Free Survival (Part A and Part B): Cervical Cancer Population
Description: Progression-free survival (PFS) was defined as the time from randomization until objective tumor progression based on response evaluation criteria in solid tumors (RECIST) version 1.1 or death. The progressive disease is defined at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. Participants who had not experienced disease progression or who were still alive at the time of evaluation were censored for the analysis. The PFS was estimated using Kaplan-Meier method.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: The objective response rate (ORR) evaluable with cervical cancer population included all participants in the All Treated Population who had cervical cancer and had at least 1 post-baseline radiologic tumor response assessment (complete response [CR], partial response [PR], stable disease [SD], or progressive disease [PD]).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part A (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736: Participants with cervical cancer received MEDI4736 3 mg/kg IV infusion Q2W at an infusion rate of approximately 60 minutes followed by ADXS11-001 1×10^9 CFU IV infusion Q4W at an infusion rate of approximately 60 minutes. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
- Part A + Part B (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736: Participants with cervical cancer received MEDI4736 10 mg/kg IV infusion Q2W at an infusion rate of approximately 60 minutes followed by ADXS11-001 1×10^9 CFU IV infusion Q4W at an infusion rate of approximately 60 minutes in Part A escalation and Part B expansion cohort. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
Arm/Group | Part A (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A + Part B (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736
Number analyzed (Participants) | 4 | 23 | 20
months | 3.7 [1.8 to 22.1] | 2.1 [1.7 to 3.8] | 5.0 [1.8 to 6.9]

3. Primary Outcome: Progression Free Survival (Part A): Human Papillomavirus (HPV)+ Head and Neck Cancer Population
Description: PFS was defined as the time from randomization until objective tumor progression based on RECIST version 1.1 or death. The progressive disease is defined at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. Participants who had not experienced disease progression or who were still alive at the time of evaluation were censored for the analysis. The PFS was estimated using Kaplan-Meier method.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: The ORR Evaluable with HPV+ head and neck cancer population included all participants in the All Treated Population who had HPV+ head and neck cancer and had at least 1 post-baseline radiologic tumor response assessment (CR, PR, SD, or PD).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part A Escalation and Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736: Participants with SCCHN received MEDI4736 10 mg/kg IV infusion Q2W at an infusion rate of approximately 60 minutes followed by ADXS11-001 1×10^9 CFU IV infusion Q4W at an infusion rate of approximately 60 minutes in Part A escalation and expansion cohorts. Treatment cycles were 8-week in duration and participants were to continue therapy for up to 1 year or until documented progression, unacceptable toxicity, withdrawal of consent, or other treatment discontinuation criteria were met.
Arm/Group | Part A Escalation and Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Number analyzed (Participants) | 12
months | 3.5 [1.6 to 5.3]

4. Primary Outcome: Percentage of Participants With Objective Response as Per RECIST Criteria (Part A and Part B): Cervical Cancer Population
Description: The objective response is defined as confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). The PR is defined as >= 30% decrease in the sum of the longest diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: ORR Evaluable with Cervical Cancer Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A + Part B (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736
Number analyzed (Participants) | 4 | 23 | 20
percentage of participants | 25.0 [0.6 to 80.6] | 8.7 [1.1 to 28.0] | 10.0 [1.2 to 31.7]

5. Primary Outcome: Percentage of Participants With Objective Response as Per RECIST Criteria (Part A): HPV+ Head and Neck Cancer Population
Description: The objective response is defined as confirmed CR or PR based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. The PR is defined as >= 30% decrease in the sum of the longest diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: ORR Evaluable with HPV+ Head and Neck Cancer Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A Escalation and Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Number analyzed (Participants) | 12
percentage of participants | 0.00 [0.0 to 0.0]

6. Primary Outcome: Percentage of Participants With Objective Response as Per irRECIST Criteria (Part A and Part B): Cervical Cancer Population
Description: The objective response is defined as confirmed CR or confirmed PR based on immune-related RECIST (irRECIST) v1.1 guidelines. The irCR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The irPR is defined as >= 30% decrease in tumor burden compared with baseline.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: ORR Evaluable with Cervical Cancer Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A + Part B (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736
Number analyzed (Participants) | 4 | 23 | 20
percentage of participants | 25.0 [0.6 to 80.6] | 8.7 [1.1 to 28.0] | 10.0 [1.2 to 31.7]

7. Primary Outcome: Percentage of Participants With Objective Response as Per irRECIST Criteria (Part A): HPV+ Head and Neck Cancer Population
Description: The objective response is defined as confirmed CR or confirmed PR based on irRECIST v1.1 guidelines. The irCR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The irPR is defined as >= 30% decrease in tumor burden compared with baseline.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: ORR Evaluable with HPV+ Head and Neck Cancer Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A Escalation and Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Number analyzed (Participants) | 12
percentage of participants | 0.00 [0.0 to 0.0]

8. Primary Outcome: Percentage of Participants With Disease Control as Per RECIST Criteria (Part A and Part B): Cervical Cancer Population
Description: The DCR is defined percentage of participants with CR, PR, or stable disease (SD) based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. The PR is defined as >= 30% decrease in the sum of the longest diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the study treatment started. The PD is defined as at least 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: ORR Evaluable with Cervical Cancer Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A + Part B (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736
Number analyzed (Participants) | 4 | 23 | 20
percentage of participants | 50.0 [6.8 to 93.2] | 47.8 [26.8 to 69.4] | 65.0 [40.8 to 84.6]

9. Primary Outcome: Percentage of Participants With Disease Control as Per RECIST Criteria (Part A): HPV+ Head and Neck Cancer Population
Description: The DCR is defined percentage of participants with CR, PR, or SD based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. The PR is defined as >= 30% decrease in the sum of the longest diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the study treatment started. The PD is defined as at least 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: ORR Evaluable with HPV+ Head and Neck Cancer Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A Escalation and Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Number analyzed (Participants) | 12
percentage of participants | 58.3 [27.7 to 84.8]

10. Primary Outcome: Percentage of Participants With Disease Control as Per irRECIST Criteria (Part A and Part B): Cervical Cancer Population
Description: The DCR is defined percentage of participants with irCR, irPR, or irSD based on irRECIST v1.1 guidelines. The irCR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The irPR is defined as >= 30% decrease in tumor burden compared with baseline. The irSD is defined as neither a 30% decrease in tumor burden compared with baseline nor a 20% increase compared with nadir can be established.
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: ORR Evaluable with Cervical Cancer Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A + Part B (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736
Number analyzed (Participants) | 4 | 23 | 20
percentage of participants | 75.0 [19.4 to 99.4] | 52.2 [30.6 to 73.2] | 65.0 [40.8 to 84.6]

11. Primary Outcome: Percentage of Participants With Disease Control as Per irRECIST Criteria (Part A): HPV+ Head and Neck Cancer Population
Description: as for outcome 10
Time Frame: From randomization until objective tumor progression or death (maximum duration: 146 weeks)
Population: ORR Evaluable with HPV+ Head and Neck Cancer Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A Escalation and Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Number analyzed (Participants) | 12
percentage of participants | 50.0 [21.1 to 78.9]

12. Primary Outcome: Overall Survival: Cervical Cancer Population
Description: Overall survival is defined as the time from the date of start of study treatment until death due to any cause. Any participant not died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive. The OS was estimated using Kaplan-Meier method.
Time Frame: From first dose until death (maximum duration: 146 weeks)
Population: All Treated Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A + Part B (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736
Number analyzed (Participants) | 5 | 30 | 27
months | NA [2.8 to NA] — Median, and upper limits of 95% CI were not estimable as more than 50% of participants were censored. | 9.3 [6.0 to NA] — Upper limits of 95% CI were not estimable as more than 50% of participants were censored. | 9.2 [6.9 to NA] — Upper limits of 95% CI were not estimable as more than 50% of participants were censored.

13. Primary Outcome: Overall Survival: HPV+ Head and Neck Cancer Population
Description: as for outcome 12
Time Frame: From first dose until death (maximum duration: 146 weeks)
Population: All Treated Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A Escalation and Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
Number analyzed (Participants) | 13
months | 4.8 [3.6 to NA] — Upper limits of 95% CI were not estimable as more than 50% of participants were censored.

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization until end of study (maximum duration: 146 weeks). Adverse events: From first dose until 30 days after last dose (maximum duration: 98 weeks)
Description: All-cause mortality: All participants who were randomized in the study. Adverse events: All Treated Population.
Arm/Group | Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 | Part A Escalation (Cervical and Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part A Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 10 mg/kg MEDI4736 | Part B Expansion (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736
All-Cause Mortality (participants affected / at risk) | 2/5 | 2/5 | 7/11 | 8/27 | 12/27
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/5 | 4/11 | 13/27 | 15/27
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 11/11 | 25/27 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 (N=5) | Part A Escalation (Cervical and Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (N=5) | Part A Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (N=11) | Part B Expansion (Cervical): 10 mg/kg MEDI4736 (N=27) | Part B Expansion (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (N=27)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestine obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 3 | 4
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Performance status decreased (General disorders) | 0 | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory track infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Metastasis to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 2
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Escalation (Cervical): 1×10^9 CFU ADXS11-001/ 3 mg/kg MEDI4736 (N=5) | Part A Escalation (Cervical and Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (N=5) | Part A Expansion (Head and Neck): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (N=11) | Part B Expansion (Cervical): 10 mg/kg MEDI4736 (N=27) | Part B Expansion (Cervical): 1×10^9 CFU ADXS11-001/ 10 mg/kg MEDI4736 (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 10 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 2 | 3 | 1 | 8
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 1 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 2
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 5 | 12
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Levator syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 4 | 12
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Tongue discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 5 | 11
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1
Chills (General disorders) | 4 | 5 | 1 | 1 | 18
Disease progression (General disorders) | 0 | 1 | 0 | 3 | 4
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 5 | 8 | 12
Influenza like illness (General disorders) | 0 | 1 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2 | 1
Oedema peripheral (General disorders) | 2 | 0 | 1 | 1 | 4
Pain (General disorders) | 0 | 0 | 0 | 0 | 3
Performance status decreased (General disorders) | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 3 | 3 | 3 | 13
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 5 | 0 | 7
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Stoma site candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 5 | 2
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 4 | 5
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 2 | 4
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 2
Po2 decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 1
Respiratory rate decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Thyroxine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Tri-iodothyronine decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 1 | 0 | 1 | 0 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 2 | 0 | 3
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 3 | 4 | 8
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 4 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 4 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 3
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 3 | 9
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 3
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 2
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 2 | 2
Embolism (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 2
Hypotension (Vascular disorders) | 1 | 2 | 5 | 1 | 12
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Based on a discussion with the FDA, a 1-year duration of the Listeria monocytogenes surveillance period was considered sufficient (instead of protocol specified 3-years period) to monitor and characterize any potential risk associated with delayed listeremia, and therefore, the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall seek the Sponsor's written approval for study results publication which shall not be unreasonably withheld. Such publication by Institution and/or Investigator may be no earlier than after a cooperative publication has been published with Sponsor or 1 year from date of completion or termination of the Study & only after review and comment by Sponsor. Institution agrees to provide Sponsor a copy of proposed publication at least 60 days prior to submission to a publisher.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT02291055/Prot_SAP_000.pdf